CLINICAL TRIAL: NCT03618290
Title: Plasma Free Fatty Acids Profile As A Diagnostic Tool For Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Sanford Health (Other)
Collaborators: University of North Dakota (Other)
Responsible Party: Sponsor
Other Study IDs: SHFASt2018
Record Dates: First submitted 2018-07-31; First posted 2018-08-07 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Stroke, Acute
Keywords: Acute ischemic stroke; plasma free fatty acid
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples in volume of 5 ml will be collected three times within a 24 hour period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute ischemic stroke group: 50 patients (expected) - Acute ischemic stroke (AIS)
  Interventions: Diagnostic Test: Analyze plasma free fatty acid in blood
- Non-neurological pathologies group: 25 control subjects with non-neurological pathologies (Congestive heart failure (CHF), Chronic obstructive pulmonary disease ( COPD ) etc.)
  Interventions: Diagnostic Test: Analyze plasma free fatty acid in blood
- Non AIS-related brain injuries group: 25 control subjects with traumatic or other non AIS-related brain injuries. These will include: Traumatic Brain Injury (TBI) defined as intracranial hemorrhage or contusion.
  Interventions: Diagnostic Test: Analyze plasma free fatty acid in blood

INTERVENTIONS:
Diagnostic Test: Analyze plasma free fatty acid in blood — This study is prospectively designed with the purpose of investigating potential new lipid targets and the free fatty acids as specific markers of acute brain injury.
  Dynamic measurement of lipid profile in 3 consecutive samples at (I) the time intervals of admission, (II) 8 hours and (III) 24 hours after admission will give the opportunity of comparison mass-spectrometric analysis of highly complex plasma samples thus reducing variability between analyzed samples and allowing precise focusing on essential lipid target changes during stroke progression.

SUMMARY:
The purpose of the research is to use plasma free fatty acid profiling as a biomarker for ischemic stroke. The plasma free acid profile will be specifically and significantly changed in early stages upon stroke onset, and correlate with the stroke volume and progression determined by imaging techniques.

DETAILED DESCRIPTION:
Ischemic stroke is the third leading cause of death and the leading cause of long-term disability in the United States. Immediate treatment can play a major role in the outcome of ischemic stroke and can help improve prognosis in many cases. One of the factors effecting immediate treatment is a rapid and accurate diagnostics of ischemic stroke.

Although imaging techniques remain to be the primary diagnostic instrumental tool, advanced imaging studies can slow management decisions and are sometimes unavailable. In addition, imaging studies often cannot discriminate between pre-existing lesions and acute or ongoing processes. Thus, additional diagnostic and prognosis tools such as plasma biomarkers will be beneficial for the early management of ischemic stroke. Importantly, the only FDA approved therapeutic treatment for ischemic stroke is tPA administration within 3-4.5 hours of stroke onset. Thus, the ideal biomarker for ischemic stroke would be readily detectible within this window for intravenous thrombolysis.

To date, the majority of potential stroke biomarkers studied are of peptide/protein nature and do not meet this requirement. One of the reasons is that hydrophilic substrates including peptides and proteins do not readily cross blood-brain barrier (BBB). Thus, brain specific peptides/proteins are unlikely to be significantly increased in plasma within the therapeutic windows of acute stroke conditions, but rather will be slowly increased during progression of stroke associated with BBB integrity loss. As a result, the most commonly utilized brain-specific protein biomarkers, including S100b and neuron specific enolase, do not increase in plasma before 10-18 hours, and do not correlate with infarct volume prior to 24 hours after injury. Many other brain-specific proteins studied have similar limitations, while proteins such as copeptin found elevated under acute stroke conditions are highly non-specific for the brain and may serve as a more general marker of physiologic stress. Another promising approach is utilization of blood gene expression analysis to identify the etiology of acute ischemic stroke. However, the timing of RNA expression measurement, as well as dynamics for RNA expression may add limitations to this approach to meet "the ideal ischemic stroke biomarker" requirement.

Alternatively, lipid biomarkers may overcome these limitations. Lipids are hydrophobic and readily cross the BBB, are very abounded accounting for about 10% of brain wet weight, have a brain specific profile, and alterations in brain lipids develop immediately upon ischemic injury. Recently, using a targeted quantification, a brain specific sphingolipid was identified as a promising biomarker for acute brain damage, demonstrating a feasibility of using lipid biomarkers to diagnose stroke.

In the current project, the investigators propose a novel approach of using plasma free fatty acid profiling as a biomarker for ischemic stroke. This novel approach is based on well documented features of brain lipid composition and metabolism under acute ischemia conditions. First, the brain has a unique signature of phospholipid fatty acid composition that is different from plasma and other tissues with one of the highest arachidonic, docosahexaenoic, and adrenic acid concentrations, that make up to 20% of fatty acids in the mammalian brain. These polyunsaturated fatty acids are mainly esterified in the sn-2 position on phospholipids and are released by a phospholipase of the A2 family. Secondly, lipids constitute more than half of the dry weight in human brain, making it the second greatest lipid containing organ in the body after adipose tissue, thus representing a significant potential source for fatty acids. Third, upon acute ischemic injury, brain phospholipases (predominantly A2 family) are immediately activated, leading to a rapid (within minutes) release of polyunsaturated fatty acids from sn-2 position from phospholipids in the free form. Because of the hydrophobicity of fatty acids, they are readily permeable for BBB and are expected to be found in plasma. Forth, dietary fatty acids are circulated in the esterified form, while released from adipose tissue free fatty acids have a different fatty acid profile, making brain free fatty acids distinguishable from other fatty acid pools in plasma.

The only FDA approved treatment for ischemic strokes is tissue plasminogen activator (tPA, also known as IV rtPA, given through an IV in the arm), administered within 3-4.5 hours of stroke onset. tPA works by dissolving the clot and improving blood flow to the part of the brain being deprived of blood flow. Although imaging techniques remain to be the primary diagnostic instrumental tool, advanced imaging studies can slow management decisions and are sometimes unavailable. In addition, imaging studies often cannot discriminate between pre-existing lesions and acute or ongoing processes. Thus, additional diagnostic and prognosis tools such as plasma biomarkers will be beneficial for the early management of ischemic stroke.

ELIGIBILITY:
This study will not involve children, neonates, pregnant women or prisoners.

Inclusion Criteria:

* Have onset of symptoms within 24-hours of presentation (AIS and Brain ?Trauma arms only).
* 18-years old and older.
* Able to offer informed consent after passing the MMSE with score ≥18 or able to obtain consent from legally authorized representative if MMSE score is ≤17.
* Participants must be admitted to the hospital and stay for at least 24 hours.
* Present with a traumatic or non AIS-related brain injury (non-AIS brain injury arm only).
* Diagnosed with non-neurological pathology (non-neurological pathology arm only).

Exclusion Criteria:

* Have onset of symptoms more than 24-hours before presentation (AIS and Brain Trauma arms).
* Less than 18-years old.
* Patients unwilling to provide consent with MMSE score of 18 or greater.
* Legally authorized representative unable or unwilling to provide consent for patients with an MMSE score of 17 or less.
* If they leave the hospital within 24 hours after being admitted.
* No longer meeting the eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Sanford Health Fargo, ND Emergency Room for AIS, non-neurological pathologies such as CHF, COPD etc., or with traumatic or other non AIS-related brain injuries. These will include: intracranial hemorrhage or brain contusions.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Correlation between lipid targets and an acute stroke incident | Through study completion, anticipated through to July 11, 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaliy Starosta, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No